CLINICAL TRIAL: NCT01232543
Title: An Open-Label Evaluation of the Adrenal Suppression Potential of Product 0405 in the Treatment of Moderate to Severe Atopic Dermatitis in Pediatric Subjects
Brief Title: Safety Study Evaluating the Adrenal Suppression Potential of Product 0405 in Pediatric Subjects With Atopic Dermatitis
Acronym: 0405-01-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0405-01-04
Record Dates: First submitted 2010-10-28; First posted 2010-11-02 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Product 0405 (Experimental): Topical Active Investigational Product 0405
  Interventions: Drug: Product 0405

INTERVENTIONS:
Drug: Product 0405 — Product 0405 will be administered topically, twice daily for 28 days.

SUMMARY:
The aim of the trial is to assess Adrenal Suppression potential when pediatric subjects are administered Product 0405 for the treatment of Atopic Dermatitis

DETAILED DESCRIPTION:
Treatment medication will be administered topically, twice a day for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Atopic Dermatitis
* Good health with the exception of Atopic Dermatitis
* Percent body surface area minimum requirements

Exclusion Criteria:

* Subjects who are pregnant, nursing, or planning a pregnancy

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the absence or presence of adrenal suppression. | 4 weeks

SECONDARY OUTCOMES:
Incidence of success based on the Investigators Static Global Assessment and the Clinical Signs and Symptoms (erythema, scaling) at the end of treatment. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Ocasio, CCRA, Study Director — Fougera Pharmaceuticals Inc.
Locations (1):
- Fougera Pharmaceuticals Inc., Melville, New York, United States